CLINICAL TRIAL: NCT02983539
Title: Detection of Circulating Tumor Cells in Patients With Metastatic Sarcomas
Brief Title: Detection of Circulating Tumor Cells in Patients With Sarcomas
Acronym: CTCS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: AC Camargo Cancer Center (Other)
Responsible Party: Principal Investigator, Ludmilla Thome Domingos Chinen, PhD, Researcher, AC Camargo Cancer Center
Other Study IDs: ACFrance
Record Dates: First submitted 2016-10-27; First posted 2016-12-06 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Leiomyosarcoma; Pleomorphic Liposarcoma; Synovial Sarcoma; Liposarcoma
Keywords: sarcomas; immunocytochemistry; circulating tumor cells
MeSH Terms: conditions — Leiomyosarcoma; Liposarcoma; Sarcoma, Synovial; Sarcoma; Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The sarcomas represent 1% of all cancers in adults, 8% in adolescents and young people, and 10% in children. Even though it is a rare cancer, it contributes to a significant loss of years of life in comparison with other types of cancer, due the fact that it affects children and young people. The diagnosis and treatment are difficult, considering the diversity and rarity of this disease. In addition, on average, more than 50% of patients with high-grade sarcoma present tumor relapse and distant recurrence is considered the main cause of death. The presence of Circulating Tumor Cells (CTCs) in the blood of patients with sarcoma may be an early marker of tumor invasion, because it is known that the CTCs circulate in the blood for months or years before the development of metastases. The CTCs can be used to monitor the response of the tumor to treatment, in order to match time, dose, and type of therapy.

Objectives: collect blood from patients with different types of sarcoma (leiomyosarcoma, synovial sarcoma, pleomorphic sarcoma and liposarcoma) in order to isolate and quantify CTCs. The investigators also have an intention to identify genes of resistance to treatment in these cells.

DETAILED DESCRIPTION:
Methodology: This is a prospective study, to be made by whole blood collection from 40 patients with different types of sarcomas (leiomyosarcoma, pleomorphic sarcoma, synovial sarcoma and liposarcoma). The collections will be made in three different moments: before the beginning of the treatment, during and at the end of this (8 mL). Blood samples will be processed and filtered on ISET system for the isolation and quantification of CTCs. Later, it will be performed immunocytochemistry (ICQ) single and/or double staining for protein assessment. The following proteins will be assessed: CD45, MRP1, MRP2 and MRP7.

Expected Results: The investigators hope that this study can show if the CTCs can be used as "liquid biopsy" in patients with leiomyosarcoma, synovium and pleomorphic sarcoma and liposarcoma.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or more;
* types of sarcomas: leiomyosarcoma, pleomorphic sarcoma, synovial sarcoma and liposarcoma.
* extension of the disease determined by physical examination and imaging;
* measurable disease by RECIST criteria (Response Evaluation Criteria in Solid Tumors);

Exclusion Criteria:

* patients who have undergone previous therapy in the last three weeks;
* patients with a history of other cancer in the past two years.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with 4 types of metastatic sarcomas: leiomyosarcoma, pleomorphic sarcoma, synovial sarcoma and liposarcoma.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2015-10; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
progression free survival | 6 months
  time to first progression until the second one

CONTACTS AND LOCATIONS:
Overall Officials: Ludmilla Chinen, PhD, Principal Investigator — AC Camargo Cancer Center
Locations (1):
- ACCamargo Cancer Center, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdallah EA, Fanelli MF, Souza E Silva V, Machado Netto MC, Gasparini Junior JL, Araujo DV, Ocea LM, Buim ME, Tariki MS, Alves Vda S, Piana de Andrade V, Dettino AL, Abdon Lopes de Mello C, Chinen LT. MRP1 expression in CTCs confers resistance to irinotecan-based chemotherapy in metastatic colorectal cancer. Int J Cancer. 2016 Aug 15;139(4):890-8. doi: 10.1002/ijc.30082. Epub 2016 Apr 28. PMID 26950035
- [Result] Chinen LT, Mello CA, Abdallah EA, Ocea LM, Buim ME, Breve NM, Gasparini JL Junior, Fanelli MF, Paterlini-Brechot P. Isolation, detection, and immunomorphological characterization of circulating tumor cells (CTCs) from patients with different types of sarcoma using isolation by size of tumor cells: a window on sarcoma-cell invasion. Onco Targets Ther. 2014 Sep 16;7:1609-17. doi: 10.2147/OTT.S62349. eCollection 2014. PMID 25258541